CLINICAL TRIAL: NCT04435600
Title: A Randomized, Active-Controlled, Efficacy Assessor-Blinded Study to Evaluate Pharmacokinetics, Safety and Efficacy of Risankizumab in Patients From 6 to Less Than 18 Years of Age With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of Subcutaneous Risankizumab Injection for Pediatric Participants With Moderate to Severe Plaque Psoriasis to Assess Change in Disease Symptoms
Acronym: OptIMMize-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: M19-977; 2023-504156-10-00 (Other: EU CT)
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Risankizumab; Ustekinumab; Psoriasis; Biologic; ABBV-066; SKYRIZI
MeSH Terms: conditions — Psoriasis | interventions — risankizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1: Risankizumab Dose A (Experimental): Participants age 12 to less than 18 receive fixed dose of risankizumab Dose A for 40 weeks.
  Interventions: Drug: Risankizumab
- Part 2: Ustekinumab Dose A/B/C then Risankizumab Dose A/B (Experimental): Participants age 12 to less than 18 will receive:
  Period A: Ustekinumab Dose A, Dose B, or Dose C based on body weight for 16 weeks (at Week 0 and Week 4).
  Period B: Risankizumab Dose A or B based on body weight for 24 weeks.
  Interventions: Drug: Risankizumab; Drug: Ustekinumab
- Part 2: Risankizumab Dose A/B (Experimental): Participants age 12 to less than 18 will receive:
  Period A: Risankizumab Dose A or B based on body weight for 16 weeks (at Week 0 and Week 4).
  Period B: Participants who respond to Risankizumab in Period A are re-randomized to continue Risankizumab Dose A or B based on body weight for up to 24 weeks or withdraw from treatment until flare.
  Period C: Participants withdrawn from treatment in Period B and experience a flare in symptoms at Week 28 or beyond are eligible for re-treatment with Risankizumab Dose A or B based on body weight for 16 weeks (at Week 0 and Week 4).
  Interventions: Drug: Risankizumab
- Part 3: Risankizumab Dose A/B (Experimental): Participants age 6 to less than 12 will receive Risankizumab Dose A or B based on body weight for 40 weeks.
  Interventions: Drug: Risankizumab
- Part 4: Risankizumab Dose A/B (Experimental): Participants age 6 to less than 12 will receive Risankizumab Dose A or B based on body weight for 40 weeks (Japan only: participants age 12 to less than 18 years will be included).
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection
  Other Names: SKYRIZI; ABBV-066
Drug: Ustekinumab — Subcutaneous Injection
  Arms: Part 2: Ustekinumab Dose A/B/C then Risankizumab Dose A/B

SUMMARY:
Psoriasis is a chronic, systemic, inflammatory disease in which skin cells build up and develop thick, red and white scaly patches on the skin. There is an unmet medical need for effective treatment in pediatric patients and this study is being done to evaluate risankizumab in pediatric participants with moderate to severe plaque psoriasis. This study will assess the change in disease symptoms.

Risankizumab is a drug being studied for the treatment for plaque psoriasis in pediatric participants. This study has 4 parts.

Part 1: Participants aged 12 < 18 will receive a fixed dose of risankizumab. Part 2: Participants aged 12 < 18 will receive;

* Period A: Risankizumab or ustekinumab based on body weight followed by;
* Period B: Risankizumab or no treatment.
* Period C: Re-treatment with risankizumab (if needed).

Part 3: Participants aged 6 < 12 will receive risankizumab based on body weight.

Part 4: Participants aged 6 < 12 will receive risankizumab based on body weight (Japan only: Participants aged 12 > 18 will receive risankizumab based on body weight).

Around 132 participants will be enrolled in approximately 50 sites worldwide.

Risankizumab and ustekinumab are given as a subcutaneous (under the skin) injection.

Parts 1, 3, and 4: Risankizumab for 40 weeks with a follow-up call 20 weeks later for a study duration of approximately 65 weeks.

Part 2:

* Period A: Risankizumab or ustekinumab for 16 weeks.
* Period B: Risankizumab or no treatment for 36 weeks.
* Period C: Re-treatment with risankizumab for 16 weeks. Follow-up call 20 weeks later for a study duration of approximately 81 weeks. Participants from each Part who meet eligibility criteria for an open-label extension (OLE) study may continue on risankizumab for 216 additional weeks.

There may be a higher burden for study participants compared to standard treatment. Participants will attend monthly visits and medical assessments will check the effect of treatment through blood tests, questionnaires, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic plaque psoriasis for at least 6 months before the Baseline Visit.
* Stable severe or moderate to severe plaque psoriasis as defined in each study part by body surface area (BSA) psoriasis involvement and scores on the Psoriasis Area and Severity Index (PASI) and Static Physician Global Assessment (sPGA).
* Candidate for systemic therapy as assessed by the investigator and meet the disease activity criteria at both the Screening and Baseline Visits per the protocol.

Exclusion Criteria:

- Concurrent clinically significant medical conditions other than the indication being studied or any other reason that the investigator determines would interfere with the participant's participation in this study, would make the participant an unsuitable candidate to receive study drug, or would put the participant at risk by participating in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (53):
- United States (21):
  - UAB Department of Dermatology /ID# 218834, Birmingham, Alabama
  - First OC Dermatology /ID# 217733, Fountain Valley, California
  - Integrative Skin Science and Research /ID# 221741, Sacramento, California
  - University of California San Diego - Rady Children's Hospital San Diego /ID# 217906, San Diego, California
  - Rybear, Inc /ID# 223164, Fort Lauderdale, Florida
  - Solutions Through Adv Rch /ID# 217936, Jacksonville, Florida
  - Olympian Clinical Research- St. Petersburg /ID# 217941, St. Petersburg, Florida
  - Advanced Clinical Research Institute /ID# 222706, Tampa, Florida
  - University Dermatology and Vein Clinic, LLC /ID# 222778, Darien, Illinois
  - Duplicate_Arlington Dermatology /ID# 217472, Rolling Meadows, Illinois
  - Duplicate_Skin Cancer and Dermatology Institute (SCDI) /ID# 221738, Reno, Nevada
  - Duplicate_Forest Hills Dermatology Group /ID# 227941, Kew Gardens, New York
  - Univ Hosp Cleveland /ID# 228483, Cleveland, Ohio
  - The Ohio State University /ID# 217808, Columbus, Ohio
  - Apex Clinical Research Center /ID# 228537, Mayfield Heights, Ohio
  - Vital Prospects Clinical Research Institute, PC /ID# 217960, Tulsa, Oklahoma
  - Medical University of South Carolina /ID# 217735, Charleston, South Carolina
  - Arlington Research Center, Inc /ID# 217471, Arlington, Texas
  - West Virginia University Hospitals /ID# 228352, Morgantown, West Virginia
  - Clinical Investigation Specialist, Inc - Kenosha /ID# 223161, Kenosha, Wisconsin
  - Wisconsin Medical Center /ID# 240005, Milwaukee, Wisconsin
- Canada (4):
  - Duplicate_Dermatology Research Institute Inc. /ID# 226172, Calgary, Alberta
  - Karma Clinical Trials /ID# 226177, St. John's, Newfoundland and Labrador
  - Hospital for Sick Children /ID# 226167, Toronto, Ontario
  - CHU Sainte-Justine /ID# 226170, Montreal, Quebec
- Germany (6):
  - Fachklinik Bad Bentheim /ID# 226014, Bad Bentheim, Lower Saxony
  - Universitaetsklinikum Bonn /ID# 228880, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 225988, Münster, North Rhine-Westphalia
  - Duplicate_Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz /ID# 225987, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 228881, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 226013, Kiel, Schleswig-Holstein
- Japan (6):
  - Nagoya City University Hospital /ID# 230830, Nagoya, Aichi-ken
  - Hiroshima University Hospital /ID# 256162, Hiroshima, Hiroshima
  - Mie University Hospital /ID# 230836, Tsu, Mie-ken
  - Kansai Medical University Hospital /ID# 231215, Hirakata-shi, Osaka
  - Duplicate_Teikyo University Hospital /ID# 255188, Itabashi-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 230575, Shinjuku-ku, Tokyo
- Poland (5):
  - High-Med Przychodnia Specjalistyczna /ID# 226060, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. F. Chopina w Rzeszowie /ID# 226116, Rzeszów, Podkarpackie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 228252, Gdansk, Pomeranian Voivodeship
  - Dermed Centrum Medyczne Sp. z o.o /ID# 226062, Lodz, Łódź Voivodeship
  - Dermoklinika Centrum Medyczne s.c. /ID# 226063, Lodz, Łódź Voivodeship
- Spain (5):
  - Hospital Sant Joan de Deu /ID# 225722, Esplugues de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 225721, Madrid
  - Hospital Universitario Infanta Leonor /ID# 225720, Madrid
  - Hospital Universitario 12 de Octubre /ID# 227860, Madrid
  - Complejo Hospitalario Universitario de Pontevedra /ID# 226061, Pontevedra
- United Kingdom (6):
  - Duplicate_Royal Devon University Healthcare NHS Foundation Trust /ID# 228078, Exeter, Devon
  - Duplicate_University Hospital Plymouth NHS Trust /ID# 227230, Plymouth, Devon
  - Guys and St Thomas NHS Foundation Trust /ID# 227224, London, Greater London
  - Chelsea and Westminster Hospital /ID# 227231, London, Greater London
  - NHS Greater Glasgow and Clyde /ID# 227226, Glasgow, Scotland
  - Frimley Health NHS Foundation Trust /ID# 229525, Camberley, Surrey

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-977

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 139 participants were sequentially enrolled in the trial. Two participants in Part 4 were excluded from the Intent To Treat (ITT) Population because they were not from the same age cohort as the population studied in Part 4 (children) but were added to Part 4 for administrative reasons (closure of Part 2 enrollment).
Groups:
- Part 1: Risankizumab; Part 3: Risankizumab; Part 4: Risankizumab: Participants received open-label risankizumab by subcutaneous injection at weeks 0, 4, 16, 28, and 40.
- Part 2 Period A: Ustekinumab: Participants received ustekinumab by subcutaneous injection at Weeks 0 and 4.
- Part 2 Period A: Risankizumab: Participants received risankizumab by subcutaneous injection at Weeks 0 and 4.
- Part 2 Period A: Ustekinumab; Period B: Risankizumab: Participants who received ustekinumab in Part 2 Period A received risankizumab by subcutaneous injection at Weeks 16, 28, and 40.
- Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab: Participants who did not respond to risankizumab in Part 2 Period A received risankizumab by subcutaneous injectionat Weeks 16, 28, and 40.
- Part 2 Period A Risankizumab Responders; Period B: Risankizumab: Participants who responded to risankizumab in Part 2 Period A received risankizumab by subcutaneous injection at Weeks 16, 28, and 40.
- Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal: Participants who responded to risankizumab in Part 2 Period A received no treatment in Part 2 Period B.
- Part 2 Period C: Risankizumab: Participants randomized to the treatment withdrawal arm in Part 2 Period B who experienced a disease flare on or after Week 28 received risankizumab by subcutaneous injection at Weeks 0 and 4 of the 16-week re-treatment period.
Period: Part 1 (Baseline to Week 40)
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 2 Period A: Ustekinumab; Period B: Risankizumab | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal | Part 2 Period C: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Started | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period A (Baseline to Week 16)
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 2 Period A: Ustekinumab; Period B: Risankizumab | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal | Part 2 Period C: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Started | 0 | 28 | 54 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 28 | 53 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period B (Week 16 to Week 52)
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 2 Period A: Ustekinumab; Period B: Risankizumab | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal | Part 2 Period C: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Started | 0 | 0 | 0 | 28 | 10 | 22 | 21 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 28 | 10 | 22 | 21 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period C (Week 52 to Week 68)
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 2 Period A: Ustekinumab; Period B: Risankizumab | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal | Part 2 Period C: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3 (Baseline to Week 52)
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 2 Period A: Ustekinumab; Period B: Risankizumab | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal | Part 2 Period C: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4 (Baseline to Week 52)
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 2 Period A: Ustekinumab; Period B: Risankizumab | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal | Part 2 Period C: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other than specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) Population included all enrolled participants in from Parts 1, 3, and 4, and all randomized participants from Part 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab | Total
Number analyzed (Participants) | 12 | 28 | 54 | 13 | 30 | 137
Age, Customized [Count of Participants; unit: Participants]
  6 to < 9 years | 0 | 0 | 0 | 3 | 10 | 13
  9 to < 12 years | 0 | 0 | 0 | 10 | 20 | 30
  12 to <15 years | 5 | 14 | 22 | 0 | 0 | 41
  15 to <18 years | 7 | 14 | 32 | 0 | 0 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 31 | 9 | 18 | 80
  Male | 5 | 13 | 23 | 4 | 12 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8 | 1 | 0 | 17
  Not Hispanic or Latino | 10 | 22 | 46 | 12 | 30 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 6 | 2 | 3 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 1 | 3 | 0 | 2 | 8
  White | 6 | 20 | 48 | 10 | 20 | 104
  More than one race | 2 | 1 | 1 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: score on a scale] — The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing the worst outcome (complete erythroderma of the severest degree).
  score on a scale | 21.43 (8.124) | 16.55 (7.229) | 16.39 (4.909) | 26.21 (9.158) | 18.59 (9.211) | 18.28 (7.716)
Static Physician Global Assessment (sPGA) Category [Count of Participants; unit: Participants] — The sPGA is the physician's current assessment of the average thickness, erythema, and scaling of all psoriatic lesions. Scores range from 0 (clear) to 4 (severe) with higher scores representing worse outcomes.
  Participants
    0 | 0 | 0 | 0 | 0 | 0 | 0
    1 | 0 | 0 | 0 | 0 | 0 | 0
    2 | 0 | 2 | 6 | 0 | 3 | 11
    3 | 0 | 25 | 42 | 2 | 23 | 92
    4 | 12 | 1 | 6 | 11 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 (Defined as at Least 75% Improvement in PASI)
Description: The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing the worst outcome (complete erythroderma of the severest degree). Data are reported for the percentage of participants achieving at least a 75% improvement in PASI.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in each part of the study (Parts 1-4)
Population: The Intent to Treat (ITT) Population included all enrolled participants from Parts 1, 3, and 4, and all randomized participants from Part 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Number analyzed (Participants) | 12 | 28 | 54 | 13 | 30
percentage of participants | 83.3 [51.6 to 97.9] | 85.7 [67.3 to 96.0] | 85.2 [72.9 to 93.4] | 92.3 [64.0 to 99.8] | 86.7 [69.3 to 96.2]

2. Primary Outcome: Percentage of Participants Achieving Static Physician's Global Assessment (sPGA) of Clear or Almost Clear (Score of 0 or 1)
Description: The sPGA is the physician's current assessment of the average thickness, erythema, and scaling of all psoriatic lesions. Scores range from 0 (clear) to 4 (severe) with higher scores representing worse outcomes. Data are reported for the percentage of participants achieving sPGA of clear (score of 0) or almost clear (score of 1).
Time Frame: At Week 16 of initial treatment in each part of the study (Parts 1-4)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Number analyzed (Participants) | 12 | 28 | 54 | 13 | 30
percentage of participants | 83.3 [51.6 to 97.9] | 75.0 [55.1 to 89.3] | 79.6 [66.5 to 89.4] | 84.6 [54.6 to 98.1] | 90.0 [73.5 to 97.9]

3. Primary Outcome: Percentage of Participants Achieving Static Physician's Global Assessment (sPGA) of Clear or Almost Clear (Score of 0 or 1) and With at Least 2 Grade Improvement From Baseline
Description: as for outcome 2
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in each part of the study (Parts 1-4)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Number analyzed (Participants) | 12 | 28 | 54 | 13 | 30
percentage of participants | 83.3 [51.6 to 97.9] | 67.9 [47.6 to 84.1] | 68.5 [54.4 to 80.5] | 84.6 [54.6 to 98.1] | 83.3 [65.3 to 94.4]

4. Secondary Outcome: Percentage of Participants Achieving PASI 90 (Defined as at Least 90% Improvement in PASI)
Description: The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing the worst outcome (complete erythroderma of the severest degree). Data are reported for the percentage of participants achieving at least a 90% improvement in PASI.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in each part of the study (Parts 1-4)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Number analyzed (Participants) | 12 | 28 | 54 | 13 | 30
percentage of participants | 83.3 [51.6 to 97.9] | 60.7 [40.6 to 78.5] | 64.8 [50.6 to 77.3] | 84.6 [54.6 to 98.1] | 76.7 [57.7 to 90.1]

5. Secondary Outcome: Percentage of Participants Achieving PASI 100 (Defined as at Least 100% Improvement in PASI)
Description: The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing the worst outcome (complete erythroderma of the severest degree). Data are reported for the percentage of participants achieving at least a 100% improvement in PASI.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in each part of the study (Parts 1-4)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Number analyzed (Participants) | 12 | 28 | 54 | 13 | 30
percentage of participants | 41.7 [15.2 to 72.3] | 17.9 [6.1 to 36.9] | 40.7 [27.6 to 55.0] | 53.8 [25.1 to 80.8] | 43.3 [25.5 to 62.6]

6. Secondary Outcome: Percentage of Participants Achieving Static Physician's Global Assessment (sPGA) of Clear or Almost Clear (0 or 1)
Description: as for outcome 2
Time Frame: Baseline (Week 0) and Week 16 of the re-treatment phase in Part 2 (Period C)
Population: The Intent to Treat (ITT) Population included all enrolled participants from Parts 1, 3, and 4, and all randomized participants from Part 2. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure in Part 2 Period C only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 8
percentage of participants
  Baseline (Week 0) | 12.5 [0.3 to 52.7]
  Week 16 | 62.5 [24.5 to 91.5]

7. Secondary Outcome: Percentage of Participants Achieving Static Physician's Global Assessment (sPGA) of Clear or Almost Clear (Score of 0 or 1) and With at Least 2 Grade Improvement From Baseline
Description: as for outcome 2
Time Frame: Baseline (Week 0) and Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 8
percentage of participants
  Baseline (Week 0) | 0.0 [0.0 to 36.9]
  Week 16 | 62.5 [24.5 to 91.5]

8. Secondary Outcome: Percentage of Participants Achieving PASI 50 (Defined as at Least 50% Improvement in PASI)
Description: The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing the worst outcome (complete erythroderma of the severest degree). Data are reported for the percentage of participants achieving at least a 50% improvement in PASI.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in each part of the study (Parts 1-4)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
Number analyzed (Participants) | 12 | 28 | 54 | 13 | 30
percentage of participants | 91.7 [61.5 to 99.8] | 92.9 [76.5 to 99.1] | 90.7 [79.7 to 96.9] | 100 [75.3 to 100.0] | 96.7 [82.8 to 99.9]

9. Secondary Outcome: Percentage of Participants Achieving PASI 50 (Defined as at Least 50% Improvement in PASI)
Description: as for outcome 8
Time Frame: Baseline (Week 0) and Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 8
percentage of participants
  Baseline (Week 0) | 75.0 [34.9 to 96.8]
  Week 16 | 87.5 [47.3 to 99.7]

10. Secondary Outcome: Percentage of Participants Achieving PASI 90 (Defined as at Least 90% Improvement in PASI)
Description: as for outcome 4
Time Frame: Baseline (Week 0) and Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 8
percentage of participants
  Baseline (Week 0) | 37.5 [8.5 to 75.5]
  Week 16 | 87.5 [47.3 to 99.7]

11. Secondary Outcome: Percentage of Participants Achieving PASI 100 (Defined as at Least 100% Improvement in PASI)
Description: as for outcome 5
Time Frame: Baseline (Week 0) and Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 8
percentage of participants
  Baseline (Week 0) | 0 [0.0 to 36.9]
  Week 16 | 25.0 [3.2 to 65.1]

12. Secondary Outcome: Percentage of Participants Achieving PASI 75 (Defined as at Least 75% Improvement in PASI)
Description: as for outcome 1
Time Frame: Baseline (Week 0) and Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 8
percentage of participants
  Baseline (Week 0) | 37.5 [8.5 to 75.5]
  Week 16 | 87.5 [47.3 to 99.7]

13. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Total Score
Description: The CDLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of dermatologic disease symptoms and treatment on quality of life (QOL). The CDLQI items include symptoms and feelings, daily activities, leisure, school, relationships, sleep, and treatment. Each item was scored on a 4-point scale: 0 = not at all; 1 = only a little; 2 = quite a lot; and 3 = very much. Item scores (0 to 3) were added to provide a total score range of 0 to 30 with higher scores representing greater impairment of QOL and worse outcomes. A negative change from baseline score indicated a reduced impairment of QOL.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in Part 2 (Period A)
Population: The Intent to Treat (ITT) Population included all enrolled participants from Parts 1, 3, and 4, and all randomized participants from Part 2. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure in Part 2 Period A only.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab
Number analyzed (Participants) | 27 | 49
score on a scale | -6.8 (0.66) | -7.4 (0.49)

14. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Total Score
Description: as for outcome 13
Time Frame: Baseline (Week 0) to Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 6
score on a scale | -7.5 (2.88)

15. Secondary Outcome: Change From Baseline in Family Dermatology Life Quality Index (FDLQI) Total Score
Description: The FDLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of dermatologic disease symptoms and treatment on Quality of Life (QOL) of family members. It consists of 10 questions that assess the impact of skin diseases on different aspects of the family member's QOL. Each item was scored on a 4-point scale: 0 = not at all; 1 = a little; 2 = quite a lot; and 3 = very much. Item scores (0 to 3) were added to provide a total score range of 0 to 30 with higher scores representing greater impairment of QOL and worse outcomes. A negative change from baseline score indicated a reduced impairment of QOL.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in Part 2 (Period A)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab
Number analyzed (Participants) | 24 | 48
score on a scale | -6.0 (0.84) | -6.9 (0.60)

16. Secondary Outcome: Change From Baseline in Family Dermatology Life Quality Index (FDLQI) Total Score
Description: as for outcome 15
Time Frame: Baseline (Week 0) to Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 6
score on a scale | -5.8 (3.29)

17. Secondary Outcome: Change From Baseline in Itch Numerical Rating Scale (Itch NRS)
Description: The itch NRS is an 11-point scale that participants complete to describe the intensity of their itch. The itch NRS scale scores varies between 0, representing "no itching" and 10, representing "worst itch imaginable" with higher scores representing worse outcomes. A negative change from baseline indicates less intense itching and better outcomes.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in Part 2 (Period A)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab
Number analyzed (Participants) | 27 | 45
score on a scale | -2.9 (0.50) | -3.8 (0.38)

18. Secondary Outcome: Change From Baseline in Itch Numerical Rating Scale (Itch NRS)
Description: as for outcome 17
Time Frame: Baseline (Week 0) to Week 16 of the re-treatment phase in Part 2 (Period C)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 2 Period C: Risankizumab
Number analyzed (Participants) | 6
score on a scale | -2.8 (1.68)

19. Secondary Outcome: Percentage of Participants Achieving >= 4-point Improvement in the Itch Numerical Rating Scale (in Participants With Baseline Score >= 4)
Description: The itch NRS is an 11-point scale that participants complete to describe the intensity of their itch within a 24-hour recall period. The itch NRS scale scores varies between 0, representing "no itching" and 10, representing "worst itch imaginable" with higher scores representing worse outcomes. Data are reported for the percentage of participants achieving >= 4 point improvement in the itch NRS in participants with a baseline itch NRS score of >=4.
Time Frame: Baseline (Week 0) to Week 16 of initial treatment in Part 2 (Period A)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Period A: Ustekinumab | Part 2 Period A: Risankizumab
Number analyzed (Participants) | 14 | 37
percentage of participants | 57.1 [28.9 to 82.3] | 64.9 [47.5 to 79.8]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection (Day 1) to the end of the study follow-up. The median time on follow-up was 385.5, 132.5, 130.5, 255.5, 252.0, 256.5, 250.0, 119.5, 385.0, and 386.0 days for arms Part 1: Risankizumab (Risa), Part 2 Period A (P2PA): Risa, P2PA: Ustekinumab (Uste), P2PB: Uste/Risa, P2PB Non-responders/Risa, P2PB Responders/Risa, P2PB Treatment Withdrawal, P2PC: Risa, P3: Risa, and P4: Risa respectively.
Description: All-cause mortality: all randomized participants. Adverse events: all participants who received at least 1 dose of study drug.
Groups:
- Part 1: Risankizumab: Participants received open-label risankizumab by subcutaneous injection on weeks 0, 4, 16, 28, and 40.
- Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab: Participants who did not respond to risankizumab in Part 2 Period A received risankizumab by subcutaneous injection at Weeks 16, 28, and 40.
Arm/Group | Part 1: Risankizumab | Part 2 Period A: Risankizumab | Part 2 Period A: Ustekinumab | Part 2 Period A: Ustekinumab; Period B: Risankizumab | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Risankizumab | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal | Part 2 Period C: Risankizumab | Part 3: Risankizumab | Part 4: Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/54 | 0/28 | 0/28 | 0/10 | 0/22 | 0/21 | 0/8 | 0/13 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/54 | 0/28 | 1/28 | 1/10 | 0/22 | 1/21 | 0/8 | 0/13 | 0/32
Other Adverse Events (participants affected / at risk) | 6/12 | 21/54 | 11/28 | 19/28 | 8/10 | 13/22 | 11/21 | 4/8 | 6/13 | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Risankizumab (N=12) | Part 2 Period A: Risankizumab (N=54) | Part 2 Period A: Ustekinumab (N=28) | Part 2 Period A: Ustekinumab; Period B: Risankizumab (N=28) | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab (N=10) | Part 2 Period A Risankizumab Responders; Period B: Risankizumab (N=22) | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal (N=21) | Part 2 Period C: Risankizumab (N=8) | Part 3: Risankizumab (N=13) | Part 4: Risankizumab (N=32)
EOSINOPHILIC OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Risankizumab (N=12) | Part 2 Period A: Risankizumab (N=54) | Part 2 Period A: Ustekinumab (N=28) | Part 2 Period A: Ustekinumab; Period B: Risankizumab (N=28) | Part 2 Period A Risankizumab Non-responders; Period B: Risankizumab (N=10) | Part 2 Period A Risankizumab Responders; Period B: Risankizumab (N=22) | Part 2 Period A Risankizumab Responders; Period B: Treatment Withdrawal (N=21) | Part 2 Period C: Risankizumab (N=8) | Part 3: Risankizumab (N=13) | Part 4: Risankizumab (N=32)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE HAEMATOMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 4 (6)
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL VAGINOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BODY TINEA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
LICE INFESTATION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 10 (17) | 4 (4) | 12 (20) | 4 (5) | 5 (9) | 2 (2) | 0 (0) | 1 (4) | 10 (16)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
SKIN CANDIDA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINEA VERSICOLOUR (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (3)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
HEADACHE (Nervous system disorders) | 2 (2) | 3 (4) | 3 (3) | 3 (8) | 0 (0) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 3 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
POST INFLAMMATORY PIGMENTATION CHANGE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT04435600/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT04435600/SAP_001.pdf